CLINICAL TRIAL: NCT01810523
Title: Comparative Effectiveness of Descriptive Versus Narrative Emergency Department Discharge Instructions for Patient Education on Unnecessary Testing for Ankle, Foot and Knee Injuries
Brief Title: Stories to Educate Patients With Ankle, Foot, and Knee Injuries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to methodological issues that require additional consideration prior to resuming the trial.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 817212
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Injury
Keywords: Acute; lower; extremity; not requiring; diagnostic; imaging
MeSH Terms: conditions — Wounds and Injuries; Disease | interventions — Narrative Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Narrative (Experimental): This arm will receive information regarding leg injuries and X-ray usage in narrative form in addition to standard of care discharge information.
  Interventions: Behavioral: Narrative
- Control (Placebo Comparator): This arm will receive a blank piece of paper in addition to the standard of care discharge information.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Narrative — Narrative form as described above.
  Arms: Narrative
Behavioral: Control — Blank piece of paper
  Arms: Control

SUMMARY:
Study will test the use of narratives on patient satisfaction and translation of an evidence-based approach to the use of X-rays for leg injuries in the Emergency Department (ED). The investigators will identify patients with foot, ankle, or knee injuries for whom X-rays are determined to not be needed. On discharge, patients will receive the current fact-based sheet or that plus a narrative explaining the work-up and treatment of these injuries. Outcomes will be assessed by a survey measuring patient satisfaction and understanding.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic knee, ankle or foot injury presenting to ED
* No indication for X-ray by Ottawa Rules criteria
* ED provider planning to discharge patient

Exclusion Criteria:

* X-ray obtained
* Need for X-ray by established Ottawa Rules criteria
* Children
* Pregnant women
* Patient to be admitted to the hospital
* Patient non-English speaking or illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 5 minutes after intervention
  To measure patient satisfaction, we will use a validated survey instrument. The survey asks patients 5 questions, which they answer by providing responses on a 5-point scale ranging from "Poor" to "Excellent." The questions include:
  1. My satisfaction with the amount of time spent with me by the person who evaluated and treated me was....
  2. The explanation I received of how my illness should be treated was...
  3. The way the health care provider treated me was...
  4. My overall satisfaction with my visit was...
  5. Your care provider determined that you did not need an X-ray for your injury. What is your level of satisfaction with that decision?

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States